CLINICAL TRIAL: NCT04413227
Title: A Phase Ⅰb Study Evaluating the Safety, Tolerability and Pharmacokinetics of Pegylated Recombinant Human Endostatin (PEG-ENDO) in Subjects With Advanced / Metastatic Non-small Cell Lung Cancer (NSCLC) or Other Solid Tumors
Brief Title: A Phase Ib Study With Pegylated Recombinant Human Endostatin in Advanced / Metastatic NSCLC or Other Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM181202-PEGENDO-102
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: NSCLC; Solid Tumor
Keywords: pegylated recombinant human endostatin (PEG-ENDO)
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-ENDO+Docetaxel (Experimental): PEG-ENDO( 1 mg/kg or 2mg/kg or 4mg/kg or 6mg/kg or 8mg/kg）+Docetaxel 75 mg/m2，once every 3 weeks at day 1
  Interventions: Drug: Pegylated Recombinant Human Endostatin（PEG-ENDO）

INTERVENTIONS:
Drug: Pegylated Recombinant Human Endostatin（PEG-ENDO） — PEG-ENDO 1 mg/kg or 2 mg/kg or 4 mg/kg or 6 mg/kg or 8 mg/kg+Docetaxel 75 mg/m2，once every 3 weeks at day 1
  Other Names: Docetaxel

SUMMARY:
The primary purpose of this study is to examine the safety, tolerability and pharmacokinetics of PEG-ENDO in combination with docetaxel in subjects previously treated or untreated (standard therapy is not suitable or without standard therapy) for advanced or metatatic non-small cell lung cancer (NSCLC) or other solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation study in subjects with advanced or metatatic non-small cell lung cancer (NSCLC) or other solid tumors.There will be five cohorts planning as following:

cohort 1: PEG-ENDO 1 mg/kg+Docetaxel 75 mg/m2,once every 3 weeks at day 1 cohort 2: PEG-ENDO 2mg/kg+Docetaxel 75 mg/m2,once every 3 weeks at day 1 cohort 3: PEG-ENDO 4 mg/kg+Docetaxel 75 mg/m2,once every 3 weeks at day 1 cohort 4: PEG-ENDO 6 mg/kg+Docetaxel75 mg/m2,once every 3 weeks at day 1 cohort 5: PEG-ENDO 8 mg/kg+Docetaxel75 mg/m2, once every 3 weeks at day 1

* Every 3 weeks as a treatment cycle. Subjects received only PEG-ENDO in the first cycle. For second cycle or the higher, they received a combination therapy of PEG-ENDO and docetaxel. Docetaxel was limited in 4 or 6 cycles。 The observation period of DLT was the 21 days after the first administration of PEG-ENDO. During the observation period of DLT (cycle 1), subjects only receive the corresponding dose of PEG-ENDO , for the second cycle and higher ,they will treated with the combination of PEG-ENDO and Docetaxel until disease progression (PD) or intolerance . Docetaxel was limited in 4 or 6 cycles。

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent.
2. 18-70years old, male or female.
3. Histological or cytological confirmation diagnosis of Non Small Cell Lung Cancer(NSCLC) or other solid tumor, previous treated with standard therapy , or standard therapy not suitabl ,or without standard therapy.
4. At least one measurable disease according to RECIST v1.1.
5. Life expectancy of at least 3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
7. Demonstrate adequate organ function -

Exclusion Criteria:

1. uncontrolled primary CNS tumors, brain metastases, or meningeal metastases.
2. Evidence of a tumor that compresses or invades major blood vessels.
3. History of hemoptysis (>1/2 teaspoon per event) or severe bleeding or evidence of bleeding disorders in the last 3 months.
4. Clinically significant active cardiovascular disease within 6 months prior to planned start of PEG-ENDO.
5. Prior treatment with anti-agiogenetic agent.
6. Pregnant female patients; breastfeeding female patients.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | First 21days for dosing（Cycle1，each cycle is 21 days)
  Incidence of Dose Limiting Toxicity
Adverse Event(AE) | From the time the subjects signed the Informed Consent Form to 28 days after the end of the study drug treatment
  Incidence of Adverse Events
Serious Adverse Event(SAE) | From the subjects signed the Informed Consent Form to 28 days after the end of the study drug treatment
  Incidence of Serious Adverse Events
Laborarory test abnormality | From the subjects signed the Informed Consent Form to 28 days after the end of the study drug treatment
  Incidence of clinically significant laboratory abnormalities
Vital signs abnormality | From the subjects signed the Informed Consent Form to 28 days after the end of the study drug treatment
  Incidence of vital signs abnormalities
Electrocardiogram(ECG) abnormality | From the subjects signed the Informed Consent Form to 28 days after the end of the study drug treatment
  Incidence of clinically significant ECG abnormalities
Serum concentration | Pharmacokinetics(PK) blood samples are collected at pre-dose, post-dose 0,1,4,8,24,48,96,168,336,480h of cycle1 and cycle5,respectively. And the pre-dose, post-dose 0h of other required cycles.
  Serum concentration of PEG-ENDO
The maximum (or peak) serum ,Cmax | Pharmacokinetics(PK) blood samples are collected at pre-dose, post-dose 0,1,4,8,24,48,96,168,336,480h of cycle1 and cycle5,respectively. And the pre-dose, post-dose 0h of other required cycles.
  Cmax of PEG-ENDO following dose concentration.
AUC | Pharmacokinetics(PK) blood samples are collected at pre-dose, post-dose 0,1,4,8,24,48,96,168,336,480h of cycle1 and cycle5,respectively. And the pre-dose, post-dose 0h of other required cycles.
  The area under the plot of serum concentration of drug (not logarithm of the concentration) against time after drug administration.
other PK parameters | Pharmacokinetics(PK) blood samples are collected at pre-dose, post-dose 0,1,4,8,24,48,96,168,336,480h of cycle1 and cycle5,respectively. And the pre-dose, post-dose 0h of other required cycles.
  The other PK parameters (if applicable).
Maximum Tolerated Dose(MTD) | First 21days for dosing（Cycle1，each cycle is 21 days)
  To determine the Maximum Tolerated Dose (MTD) of PEG-ENDO in subjects with Advanced / Metastatic NSCLC or Other Solid Tumors

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | at least 12 weeks
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Duration of Response(DOR) | Estimated at 4 months after fist documented PD or CR
  DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1
Progression-free survival (PFS) | Estimated at 4 months.
  PFS is defined as time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by by Investigator assessment in accordance to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Huang Dingzhi, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Li Lin, Ph.D, Principal Investigator — Beijing Hospital
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Tianjin medical university cancer institute&hospital, Tianjin, Tianjin Municipality